CLINICAL TRIAL: NCT01592994
Title: Enhancing HIV Risk Reduction Among Indian Women With Risky Husbands
Acronym: RHANI Wives
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Indian Council of Medical Research (Other Government); Population Council (Other)
Responsible Party: Principal Investigator, Anita Raj, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21MH085312 (NIH)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Behavioral Risk for HIV
Keywords: HIV; condom use; India; women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): control participants received basic messages on the utility of condoms in protecting from HIV and other STIs, and they were informed about local HIV/STI counseling and testing services.
- RHANI Wives Intervention (Experimental): The RHANI Wives intervention included four household individual sessions and two small group community sessions delivered over 6-9 weeks. The intervention was based on Social Cognitive Theory (SCT) and the Theory of Gender and Power (TGP). SCT application supported focus on HIV/STI knowledge and condom skills building, as well as safer sex social norms and motivation. TGP guided the intervention focus on problem solving and skills building toward marital communication; embedded in this was gender equity counseling and support. The TGP approach allowed women to take a more active and assertive stance with husbands. Group sessions reinforced individual session knowledge and skills building and provided local social support.
  Interventions: Behavioral: RHANI WIves

INTERVENTIONS:
Behavioral: RHANI WIves — The RHANI Wives intervention included four household individual sessions and two small group community sessions delivered over 6-9 weeks. The intervention was based on Social Cognitive Theory (SCT)10 and the Theory of Gender and Power (TGP). SCT application supported focus on HIV/STI knowledge and condom skills building, as well as safer sex social norms and motivation. TGP guided the intervention focus on problem solving and skills building toward marital communication; embedded in this was gender equity counseling and support. The TGP approach allowed women to take a more active and assertive stance with husbands. Group sessions reinforced individual session knowledge and skills building and provided local social support.
  Arms: RHANI Wives Intervention

SUMMARY:
This grant involved the development, implementation, and assessment of the feasibility and acceptability of an HIV prevention intervention for at-risk wives in Mumbai, RHANI Wives (Raising HIV Awareness among Non-Infected Indian Wives). The RHANI Wives intervention was adapted from the HIV Intervention Program (HIV-IP), a community-based, multi-session HIV intervention with demonstrated effectiveness among Latinas whose primary risk for HIV was from their primary male partner (Raj et al. 2001).

Specific aims of this study are as follows:

1. To adapt HIV-IP, a culture and gender-tailored HIV intervention for Latinas with demonstrated effectiveness in reducing risk for HIV, and to create RHANI Wives for use with at-risk Indian wives.
2. To determine the feasibility and acceptability of RHANI Wives with at risk wives* in India. A two-group cluster randomized trial will involve random assignment of 12 neighborhood clusters (25 women/cluster) to receive the intervention (n=150) or a control condition (n=150). Intervention effects on the more proximal and likely safer sex mediating outcome of marital communication for this feasibility trial will be assessed via surveys at baseline and 3 month follow-up.

NOTE: Only 220 participants were able to be recruited into the study.

*At risk wives are defined as having a husband at higher risk for transactional sex based on wife's reports of his risky alcohol use (drunk in past 30 days, 3+ drinking days in past 7 days) or partner violence perpetration

ELIGIBILITY:
Inclusion Criteria:

1. married female aged 18-40 years
2. fluency in Hindi or Marathi
3. residence with husband in the area of study for a period of 2 months or greater
4. reports that husband engaged in either heavy drinking- past 30 day drunken behavior, or frequent drinking- 3 drinking days in past 7 days, or lifetime spousal violence perpetration
5. no plans to relocate from the area in the next year.

Exclusion Criteria:

* cognitive impairment indicated at recruitment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
condom use | 4.5 months
  condom protected sex in marital relationships

CONTACTS AND LOCATIONS:
Overall Officials: Anita Raj, PhD, Principal Investigator — UCSD Division of Global Public Health
Locations (1):
- Community, Bhāndup, Mumbai, India

REFERENCES:
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505
- [Derived] Saggurti N, Nair S, Silverman JG, Naik DD, Battala M, Dasgupta A, Balaiah D, Raj A. Impact of the RHANI Wives intervention on marital conflict and sexual coercion. Int J Gynaecol Obstet. 2014 Jul;126(1):18-22. doi: 10.1016/j.ijgo.2014.01.015. Epub 2014 Apr 3. PMID 24795094